CLINICAL TRIAL: NCT00359684
Title: Use of Cysteamine in the Treatment of Cystinosis
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 780093; 78-HG-0093
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-04-08

CONDITIONS: Cystinosis
Keywords: Cystinosis; Cystine; Lysomal Storage Disease; Mutation Analysis; Metabolic Disease; Natural History
MeSH Terms: conditions — Cystinosis; Metabolic Diseases | interventions — Cysteamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cystinosis: Patients with a diagnosis of cystinosis
  Interventions: Drug: Cysteamine

INTERVENTIONS:
Drug: Cysteamine — Cystine-depleting agent

SUMMARY:
Cystinosis is an inherited disease resulting in poor growth and kidney failure. There is no known cure for cystinosis, although kidney transplantation may help the renal failure and prolong survival. Both the kidney damage and growth failure are thought to be due to the accumulation of the amino acid cystine within the cells of the body. The cystine storage later damages other organs besides the kidneys, including the thyroid gland, pancreas, eyes, and muscle.

The drug cysteamine (Cystagon; ProCysBi) is an oral medication given to patients with cystinosis prior to kidney transplantation. The drug works by reducing the level of cystine in the white blood cells and muscle tissue. The drug may also decrease levels of cystine in the kidneys and other tissues.

This study has several goals:

1. Long-term surveillance of cysteamine treated patients.
2. Detection of new non-kidney complications of cystinosis.
3. Maintenance of a patient population for genetic testing (mutational analysis) of the cystinosis gene.<TAB>

   ...

DETAILED DESCRIPTION:
Patients with nephropathic cystinosis have been treated with the cystine-depleting agent cysteamine since 1978. This therapy prevents or delays renal deterioration, improves growth, and depletes parenchymal tissues of cystine. Based largely upon data produced through this protocol, the Food and Drug Administration approved cysteamine bitartrate for use in cystinosis patients on August 15, 1994. Cysteamine is available as CystagonR through Mylan Pharmaceuticals in 50 mg and 150 mg capsules and as ProcysbiR in 75 mg capsules. By virtue of the current protocol, patients are admitted to the NIH Clinical Center for investigations every two years, except for cases of great interest or urgency. On each 1-3 day admission, a battery of tests is performed and the adequacy of cystine depletion by cysteamine is monitored. This protocol demonstrates the course of cystinosis patients treated with cysteamine, describes new complications of the disorder in poorly treated adults, and maintains NHGRI expertise in the field. Its monitoring and followup of patients over the course of 3 decades represents an invaluable contribution to our understanding of the natural history of this rare disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of cystinosis, whether classical or one of the variants with later onset or no renal complications.

Patients will be diagnosed as having cystinosis based upon a leucocyte cystine content greater than 1 nmol half-cystine/mg protein (normal, less than 0.2) and a typical clinical course.

EXCLUSION CRITERIA:

Inability to travel to the NIH.

Age less than one week.

Nonviable neonates and neonates of uncertain viability will be excluded.

Ages: 1 Week to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of cystinosis
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 1979-01-04 (Actual)

PRIMARY OUTCOMES:
Serve as a source of knowledge and advice for individual cystinosis patients and for the community at large | Follow-up can occur every two years
  Serve as a source of knowledge and advice for individual cystinosis patients and for the community at large

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
pending
Supporting Information: Study Protocol
Time Frame: pending
Access Criteria: pending

REFERENCES:
- [Background] Florenzano P, Ferreira C, Nesterova G, Roberts MS, Tella SH, de Castro LF, Brown SM, Whitaker A, Pereira RC, Bulas D, Gafni RI, Salusky IB, Gahl WA, Collins MT. Skeletal Consequences of Nephropathic Cystinosis. J Bone Miner Res. 2018 Oct;33(10):1870-1880. doi: 10.1002/jbmr.3522. Epub 2018 Jul 20. PMID 29905968
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1978-HG-0093.html